CLINICAL TRIAL: NCT04647565
Title: Alcohol and Women : Screening in General Medicine.
Brief Title: Alcohol and Women : Screening in General
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0611
Record Dates: First submitted 2020-11-23; First posted 2020-12-01 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Alcoholism
Keywords: women reporting alcohol abuse and/or dependence; women recruted during hospitalisation and/or consultation; Alcohol
MeSH Terms: conditions — Alcoholism | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: interviews — interviews (human and social sciences)

SUMMARY:
The alcohol consumption of adults has been decreasing in France since the sixties. When focusing on the particular case of women, this trend goes on the opposite direction. In addition, the impact of drinking alcohol involves an increased severity in women in comparison to men. Furthermore, women consult less often doctors about their alcohol problem due to stigmatisation. Finally, as alcohol consumption is a major public health issue (second preventable cause of death), the aim of this study is to propose an earlier screening of women with alcohol use disorders (AUD) in general medicine.

DETAILED DESCRIPTION:
To improve the screening of women with AUD in general médicine, from their perceptions and experiences, and to create a screening tool to general practitioners.

The chosen method is a qualtitative study through semi-structured interview with women with AUD.

A qualitative assessment of these individual interviews could show various topics.

ELIGIBILITY:
Inclusion criteria:

- over 18 years old alcoholic women, with one or several addiction, from all social class.

Exclusion criteria:

- not being able to answer the questionnaire

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Over 18 years old alcoholic womens, medical caring in consultation with addictologist or in hospitalisation for withdrawal.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Assessment of women's opinion on an alcoholism screening by general practitioners. | 1 year
  Assessment of women's opinion on an alcoholism screening by general practitioners : Qualitative study based on semi-structured interview with women with AUD.
Creation of a screening tool dedicated to general practitioners | 1 year
  Creation of a screening tool dedicated to general practitioners : Built of a screening tool based both on litterature review about alcohol & women and a qualitative study on women's opinion.

CONTACTS AND LOCATIONS:
Overall Officials: Claire MONTADE, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC